CLINICAL TRIAL: NCT01320163
Title: Clinical Acceptability of I-GEL® in Pediatric Patients: Comparison of Clinical Performance With Classic-LMA™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assisstant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1001-019-306
Record Dates: First submitted 2011-03-17; First posted 2011-03-22 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: i-gel airway (Intersurgical Ltd., Wokingham, England) — supra-glottic airway device
Device: Laryngeal Mask Airway — supra-glottic airway device

SUMMARY:
This study is designed to determine whether a functional difference exists between the laryngeal mask airway (LMA)-Classic™ and i-gel in anesthetized children who have received neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, Mallampati I or II, presenting for elective surgery who require general anesthesia in whom tracheal intubation is not necessary

Exclusion Criteria:

* Patients will be excluded from the study if they present as Mallampati III or IV, ASA III-V or emergency status
* upper airway abnormality

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
airway leak pressure | within 5 min of insertion of each device
  Airway leak pressure was determined by adjusting the expiratory valve of the breathing circle to 40 cmH2O (fixed fresh gas flow 3 L/min) and recording the pressure when equilibrium was reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea